CLINICAL TRIAL: NCT05195138
Title: Mindfulness-Based Diabetes Education for Adults With Elevated Diabetes Distress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Caroline Presley, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300008617
Record Dates: First submitted 2021-12-23; First posted 2022-01-18 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes distress; Mindfulness-based diabetes education
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Diabetes Education (Experimental): Mindfulness-Based Diabetes Education (MBDE) will be delivered in-person in a group of 10-14 participants during 8 weekly sessions followed by 2 bimonthly individual sessions. Sessions integrate Mindfulness-Based Stress Reduction and Diabetes Self-Management Education. MBDE will introduce breath awareness meditation, body scan, walking meditation, mindful yoga, and applying mindfulness to daily activities, as well as core areas from DSME. MBDE will include incremental goal setting to build participants' self-efficacy for diabetes self-management behaviors, mindful attention to diabetes self-management, and on development of social support in the group. Participants will complete daily home mindfulness exercises and self-monitoring of diabetes self-management behaviors.
  Interventions: Behavioral: Mindfulness-Based Diabetes Education
- Standard Diabetes Self-Management Education (Active Comparator): Standard DSME will be delivered in-person, in a group setting with 10-14 participants per group. Standard DSME will be delivered by a certified diabetes educator in eight weekly sessions of 2 hours duration. Sessions will cover seven core content areas - healthy eating, physical activity, medication usage, self-monitoring, preventing and treating acute and chronic complications, healthy coping, and problem solving.
  Interventions: Behavioral: Standard Diabetes Self-Management Education (DSME)

INTERVENTIONS:
Behavioral: Mindfulness-Based Diabetes Education — Mindfulness-Based Diabetes Education described in study arm.
  Arms: Mindfulness-Based Diabetes Education
Behavioral: Standard Diabetes Self-Management Education (DSME) — Standard DSME described in study arm.
  Arms: Standard Diabetes Self-Management Education

SUMMARY:
Diabetes distress is common affecting over one-third of people with type 2 diabetes, negatively impacting self-management and outcomes, and disproportionately affecting low-income individuals. The proposed project will conduct a pilot randomized controlled trial comparing Mindfulness-Based Diabetes Education to standard Diabetes Self-Management Education in adults with type 2 diabetes and elevated diabetes distress who receive care within safety-net healthcare systems in order to assess feasibility and acceptability.

DETAILED DESCRIPTION:
The investigators will conduct a pilot randomized controlled trial (RCT) of Mindfulness-Based Diabetes Education (MBDE) versus standard Diabetes Self-Management Education (DSME) in adults with type 2 diabetes and moderate-severe diabetes distress who receive their care from safety-net healthcare systems. The goal of this pilot RCT will be to assess the acceptability and feasibility of MBDE; acceptability will be assessed through qualitative follow-up interviews with participants and feasibility will be assessed through process measures. The investigators will recruit up to approximately 96 participants, 48 from each site to account for potential loss to follow up of up to 20%, for the study with total study duration of 6 months. Participants will be randomized 1:1 to each study arm. This study will also serve as a pilot test for the procedures of the RCT and of measures to be used in participant assessments.

The study will be conducted at two safety-net clinics that provide care for residents of Jefferson County using a sliding scale program based on income level - Cooper Green Mercy Health Services Authority (CGMHSA) and Alabama Regional Medicine Services (ARMS). CGMHSA, an affiliate of University of Alabama at Birmingham (UAB) Health System, is Jefferson County's public safety-net health care facility. CGMHSA provides care primarily to the indigent county residents, geographically spanning most of the Birmingham metropolitan area. Ambulatory care services are provided to patients who have type 2 diabetes through Cooper Green's Primary Care Clinic and multi-disciplinary Diabetes Clinic. ARMS is a Community Health Center serving the greater Birmingham area since 1983. ARMS provides ambulatory care for adults, including primary care, diabetes self-management education classes, and behavioral health services. ARMS offers services to patients, with or without insurance, on a sliding scale fee program based on income.

Trained study staff overseen by the study PI will recruit participants from CGMHSA and ARMS through three methods. Opt-out letters will be mailed to patients seen at CGMHSA or ARMS in the preceding three years with a diagnosis of type 2 diabetes; study staff will then call potential participants to provide more information about the study and to gauge their interest in participating. The investigators will obtain a HIPAA waiver to access potential participant information from the medical record in order to generate a recruitment list. The investigators will also conduct in-person recruitment of participants at CGMHSA and ARMS, as well as direct referral of potential participants by providers or patients. Trained study personnel will obtain screening consent from potential participants prior to screening for eligibility based on inclusion and exclusion criteria, which will include assessment of diabetes distress and hemoglobin A1c (A1C) through point-of-care (POC) finger-stick sample. Study staff will then obtain informed consent from eligible participants at the time of enrollment.

Both MDBE and standard DSME study arms will be delivered in-person, in a group setting with 10-14 participants per group. MBDE will be delivered in 8 weekly group sessions followed by 2 bimonthly individual, booster sessions conducted by phone for a total duration of 6 months. MBDE will be delivered by an interventionist with a background in nursing and training as an MBSR instructor, who will receive additional training in MBDE with an emphasis on content drawn from DSME. Standard DSME will be delivered by a certified diabetes educator in eight weekly sessions of 2 hours duration. Sessions will cover seven core content areas - healthy eating, physical activity, medication usage, self-monitoring, preventing and treating acute and chronic complications, healthy coping, and problem solving.

Total study duration will be six months; a trained study staff will complete assessments of participants in both study arms at baseline, 2 months, and 6 months. Participants in both study arms will complete assessments that will be conducted by trained study personnel, including interviewer-administered questionnaire, biometric assessment (height, weight, blood pressure), and POC A1C testing from a finger-stick sample at 3 time points - baseline, 2 months, and 6 months. Participants in the MBDE arm will be asked to participate in a focus group (estimated length 1 hour) at the 2 month time point. Participants will receive an incentive for their participation for each study assessment and for participation in a focus group.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19-70 years
2. Diagnosis of type 2 diabetes (based on the presence of two or more outpatient International Classification of Diseases (ICD-10) codes for type 2 diabetes
3. Receipt of care at Cooper Green Mercy Health Systems Authority or Alabama Regional Medical Services (one or more visits to primary care or diabetes clinic within the prior year
4. Presence of moderate-severe diabetes distress (score ≥2 on Diabetes Distress Scale
5. Suboptimal glycemic control (elevated hemoglobin A1c (A1C) ≥7.5%)

Exclusion Criteria:

1. Non-English speaking
2. Currently pregnant
3. Diagnosis of severe psychiatric comorbidity including bipolar disorder, schizophrenia, or a history of psychosis (based on participant self-report)

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Participant assessment of perceived positive and negative effects | 2 months
  Will be assessed through focus groups with participants after they have completed the 8-weekly intervention sessions for MBDE. Interviews will be recorded and transcribed. A combined inductive/deductive approach will be used for qualitative analysis, to identify themes reported by participants.
Participant assessment of intervention content | 2 months
  Will be assessed through focus groups with participants after they have completed the 8-weekly intervention sessions for MBDE. Interviews will be recorded and transcribed. A combined inductive/deductive approach will be used for qualitative analysis, to identify themes reported by participants.
Participant assessment of appropriateness of intervention duration and frequency | 2 months
  Will be assessed through focus groups with participants after they have completed the 8-weekly intervention sessions for MBDE. Interviews will be recorded and transcribed. A combined inductive/deductive approach will be used for qualitative analysis, to identify themes reported by participants.
Participant satisfaction with interventionist | 2 months
  Will be assessed through focus groups with participants after they have completed the 8-weekly intervention sessions for MBDE. Interviews will be recorded and transcribed. A combined inductive/deductive approach will be used for qualitative analysis, to identify themes reported by participants.
Participant-reported barriers to engagement with the intervention sessions or content | 2 months
  Will be assessed through focus groups with participants after they have completed the 8-weekly intervention sessions for MBDE. Interviews will be recorded and transcribed. A combined inductive/deductive approach will be used for qualitative analysis, to identify themes reported by participants.
Participants' suggestions to improve the intervention | 2 months
  Will be assessed through focus groups with participants after they have completed the 8-weekly intervention sessions for MBDE. Interviews will be recorded and transcribed. A combined inductive/deductive approach will be used for qualitative analysis, to identify themes reported by participants.
Participants' overall satisfaction with the intervention | 2 months
  Will be assessed through focus groups with participants after they have completed the 8-weekly intervention sessions for MBDE. Interviews will be recorded and transcribed. A combined inductive/deductive approach will be used for qualitative analysis, to identify themes reported by participants.
Feasibility: percentage of screened participants who are eligible | 6 months
  We will assess the percentage of screened participants who are eligible to participate in the study. Study staff will track the number of participants who are screened for participation and the number of participants who are eligible to participate.
Feasibility: percentage of eligible participants who enroll | 6 months
  We will assess the percentage of eligible participants who enroll in the study. Study staff will track the number of participants who are eligible for participation and the number of participants who enroll in the study.
Feasibility: ability to randomize participants to study arms | 6 months
  We will assess the percentage of eligible participants who are randomized. Study staff will track the number of participants who are enrolled and the number of participants who are randomized.
Feasibility: distribution of participants by demographics | 6 months
  We will collect demographics of study participants, including age, race, ethnicity, and gender by participant self-report. This information will be obtained during a questionnaire administered to participants in English by a trained interviewer. We will use descriptive statistics to characterize the demographics of the study sample.
Feasibility: percentage of sessions attended | 6 months
  We will track the number of sessions attended by each participant and calculate the percentage of sessions attended by each participant.
Feasibility: participant adherence to study tasks include home mindfulness practices, self-monitoring activities | 6 months
  At each session, we will collect logs of participants' home mindfulness and self-monitoring activities. We will calculate participant adherence to recommended activities for each participant.
Feasibility: barriers to participation in intervention sessions or completing study activities at home | 6 months
  We will collect information from participants to assess any barriers they experienced attending study sessions or completing recommended home activities. This information will be obtained during a questionnaire administered to participants in English by a trained interviewer.
Feasibility: reasons for dropping out | 6 months
  We will collect information from participants who drop out of the intervention or study regarding the reason for dropping out.
Feasibility: overall study retention | 6 months
  We will track the number of participants who enroll in the study and complete assessments at each time point - baseline, 2 months, and 6 months.

SECONDARY OUTCOMES:
Hemoglobin A1c | Baseline
  Participants will have a point-of-care A1C measured; A1C will be obtained by trained study personnel using finger-stick testing with the A1C NOW+ Test Kits (PTS Diagnostics). A1C reports a % glycated hemoglobin level; a higher score indicates higher average blood glucose levels over the preceding 3 months. An A1C greater than or equal to 7.5% indicates poorly controlled type 2 diabetes.
Hemoglobin A1c | 6 months
  Participants will have a point-of-care A1C measured; A1C will be obtained by trained study personnel using finger-stick testing with the A1C NOW+ Test Kits (PTS Diagnostics). A1C reports a % glycated hemoglobin level; a higher score indicates higher average blood glucose levels over the preceding 3 months. An A1C greater than or equal to 7.5% indicates poorly controlled type 2 diabetes.
Diabetes distress | Baseline
  Participants will complete the Diabetes Distress Scale (DDS), a 17-item self-report measure, assessing domains of emotional burden, physician-related distress, regimen-related distress, and interpersonal distress. The mean item score yields a possible score from 1 to 6; a score of <2 indicates little/no distress, 2 to 2.9 moderate distress, and ≥3 high distress. The questionnaire will be administered to participants in English by a trained interviewer.
Diabetes distress | 2 months
  Participants will complete the Diabetes Distress Scale (DDS), a 17-item self-report measure, assessing domains of emotional burden, physician-related distress, regimen-related distress, and interpersonal distress. The mean item score yields a possible score from 1 to 6; a score of <2 indicates little/no distress, 2 to 2.9 moderate distress, and ≥3 high distress. The questionnaire will be administered to participants in English by a trained interviewer.
Diabetes distress | 6 months
  Participants will complete the Diabetes Distress Scale (DDS), a 17-item self-report measure, assessing domains of emotional burden, physician-related distress, regimen-related distress, and interpersonal distress. The mean item score yields a possible score from 1 to 6; a score of <2 indicates little/no distress, 2 to 2.9 moderate distress, and ≥3 high distress. The questionnaire will be administered to participants in English by a trained interviewer.
Diabetes self-management behaviors | Baseline
  Participants will complete the Diabetes Self-Management Questionnaire, a 16-item self-report measure that assesses dietary control, blood glucose monitoring, physical activity, and healthcare use. Participants respond on a 4-point Likert scale from 0 "does not apply to me" to 3 "applies to me very much" referring to the preceding 8 weeks. Responses are summed and transformed to a 10-point scale with a higher score indicating higher adherence to the score. The questionnaire will be administered to participants in English by a trained interviewer.
Diabetes self-management behaviors | 2 months
  Participants will complete the Diabetes Self-Management Questionnaire, a 16-item self-report measure that assesses dietary control, blood glucose monitoring, physical activity, and healthcare use. Participants respond on a 4-point Likert scale from 0 "does not apply to me" to 3 "applies to me very much" referring to the preceding 8 weeks. Responses are summed and transformed to a 10-point scale with a higher score indicating higher adherence to the score. The questionnaire will be administered to participants in English by a trained interviewer.
Diabetes self-management behaviors | 6 months
  Participants will complete the Diabetes Self-Management Questionnaire, a 16-item self-report measure that assesses dietary control, blood glucose monitoring, physical activity, and healthcare use. Participants respond on a 4-point Likert scale from 0 "does not apply to me" to 3 "applies to me very much" referring to the preceding 8 weeks. Responses are summed and transformed to a 10-point scale with a higher score indicating higher adherence to the score. The questionnaire will be administered to participants in English by a trained interviewer.
Medication adherence | Baseline
  Participants will complete the Adherence to Refills and Medications-Diabetes (ARMS-D), an 11-item self-report measure that includes medication-taking and refill subscales. Example item is "How often do you forget to take your diabetes medicine(s)?" Participants respond on a 4-point Likert scale from 1 "none of the time" to 4 "all of the time." Item responses are summed, combining subscales to yield a score from 11-44 (higher scores indicate greater difficulty with medication adherence). The questionnaire will be administered to participants in English by a trained interviewer.
Medication adherence | 2 months
  Participants will complete the Adherence to Refills and Medications-Diabetes (ARMS-D), an 11-item self-report measure that includes medication-taking and refill subscales. Example item is "How often do you forget to take your diabetes medicine(s)?" Participants respond on a 4-point Likert scale from 1 "none of the time" to 4 "all of the time." Item responses are summed, combining subscales to yield a score from 11-44 (higher scores indicate greater difficulty with medication adherence). The questionnaire will be administered to participants in English by a trained interviewer.
Medication adherence | 6 months
  Participants will complete the Adherence to Refills and Medications-Diabetes (ARMS-D), an 11-item self-report measure that includes medication-taking and refill subscales. Example item is "How often do you forget to take your diabetes medicine(s)?" Participants respond on a 4-point Likert scale from 1 "none of the time" to 4 "all of the time." Item responses are summed, combining subscales to yield a score from 11-44 (higher scores indicate greater difficulty with medication adherence). The questionnaire will be administered to participants in English by a trained interviewer.
Mindfulness | Baseline
  Participants will complete the Five Facet Mindfulness Questionnaire (FFMQ), a 15-item self-report measure that assesses facets of observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Participants respond on a 5-point Likert scale from 1 "never or very rarely true" to 5 "very often or always true." Responses are summed, facet scores range from 3-15 with a higher score indicating higher levels of mindfulness.
Mindfulness | 2 months
  Participants will complete the Five Facet Mindfulness Questionnaire (FFMQ), a 15-item self-report measure that assesses facets of observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Participants respond on a 5-point Likert scale from 1 "never or very rarely true" to 5 "very often or always true." Responses are summed, facet scores range from 3-15 with a higher score indicating higher levels of mindfulness.
Mindfulness | 6 months
  Participants will complete the Five Facet Mindfulness Questionnaire (FFMQ), a 15-item self-report measure that assesses facets of observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Participants respond on a 5-point Likert scale from 1 "never or very rarely true" to 5 "very often or always true." Responses are summed, facet scores range from 3-15 with a higher score indicating higher levels of mindfulness.
Emotion regulation | Baseline
  Participants will complete the Difficulties in Emotion Regulation Scale (DERS), an 18-item self-report measure that includes subscales on awareness, clarity, goals, impulse, nonacceptance, and strategy. Participants respond on a 5-point Likert scale from 1 "almost never" to 5 "almost always." Item responses are summed, into subscale and total scales; total scores can range from 18-90 (higher score indicates more difficulty with emotion regulation). The questionnaire will be administered to participants in English by a trained interviewer.
Emotion regulation | 2 months
  Participants will complete the Difficulties in Emotion Regulation Scale (DERS), an 18-item self-report measure that includes subscales on awareness, clarity, goals, impulse, nonacceptance, and strategy. Participants respond on a 5-point Likert scale from 1 "almost never" to 5 "almost always." Item responses are summed, into subscale and total scales; total scores can range from 18-90 (higher score indicates more difficulty with emotion regulation). The questionnaire will be administered to participants in English by a trained interviewer.
Emotion regulation | 6 months
  Participants will complete the Difficulties in Emotion Regulation Scale (DERS), an 18-item self-report measure that includes subscales on awareness, clarity, goals, impulse, nonacceptance, and strategy. Participants respond on a 5-point Likert scale from 1 "almost never" to 5 "almost always." Item responses are summed, into subscale and total scales; total scores can range from 18-90 (higher score indicates more difficulty with emotion regulation). The questionnaire will be administered to participants in English by a trained interviewer.
Self-awareness | Baseline
  Participants will complete the Multidimensional Assessment of Interoceptive Awareness, a 37-item self-report measure that includes subscales on noticing, not-distracting, not-worrying, attention regulation, emotional awareness, self-regulation, body listening, and trusting. Participants respond of a 6-point Likert scale from 0 "never to 5 "always." Mean item scores for each subscale are obtained. The questionnaire will be administered to participants in English by a trained interviewer.
Self-awareness | 2 months
  Participants will complete the Multidimensional Assessment of Interoceptive Awareness, a 37-item self-report measure that includes subscales on noticing, not-distracting, not-worrying, attention regulation, emotional awareness, self-regulation, body listening, and trusting. Participants respond of a 6-point Likert scale from 0 "never to 5 "always." Mean item scores for each subscale are obtained. The questionnaire will be administered to participants in English by a trained interviewer.
Self-awareness | 6 months
  Participants will complete the Multidimensional Assessment of Interoceptive Awareness, a 37-item self-report measure that includes subscales on noticing, not-distracting, not-worrying, attention regulation, emotional awareness, self-regulation, body listening, and trusting. Participants respond of a 6-point Likert scale from 0 "never to 5 "always." Mean item scores for each subscale are obtained. The questionnaire will be administered to participants in English by a trained interviewer.
Self-efficacy as assessed by the Perceived Diabetes Self-Management Scale (PDSMS) | Baseline
  Participants will complete the PDSMS, an 8-item self-report measure that assesses the degree to which participants feel confident to perform their diabetes self-management behaviors. Participants respond on a 5-point Likert scale from 1 "strongly disagree" to 5 "strongly agree." Items are summed; possible scores range from 8 to 40, with higher scores indicating more confidence in self-managing one's diabetes. The questionnaire will be administered to participants in English by a trained interviewer.
Self-efficacy as assessed by the Perceived Diabetes Self-Management Scale (PDSMS) | 2 months
  Participants will complete the PDSMS, an 8-item self-report measure that assesses the degree to which participants feel confident to perform their diabetes self-management behaviors. Participants respond on a 5-point Likert scale from 1 "strongly disagree" to 5 "strongly agree." Items are summed; possible scores range from 8 to 40, with higher scores indicating more confidence in self-managing one's diabetes. The questionnaire will be administered to participants in English by a trained interviewer.
Self-efficacy as assessed by the Perceived Diabetes Self-Management Scale (PDSMS) | 6 months
  Participants will complete the PDSMS, an 8-item self-report measure that assesses the degree to which participants feel confident to perform their diabetes self-management behaviors. Participants respond on a 5-point Likert scale from 1 "strongly disagree" to 5 "strongly agree." Items are summed; possible scores range from 8 to 40, with higher scores indicating more confidence in self-managing one's diabetes. The questionnaire will be administered to participants in English by a trained interviewer.
Social support | Baseline
  Participants will complete the 6-item Social Support Questionnaire. For each item, respondents first list the number of individuals available for support in specific circumstances, and then indicate their level of satisfaction with that support using a 6-point Likert-type scale from 1 "dissatisfied" to 6 "very satisfied." The means of the two parts are obtained separately to indicate mean number of social supports and mean satisfaction with social support. The questionnaire will be administered to participants in English by a trained interviewer.
Social support | 2 months
  Participants will complete the 6-item Social Support Questionnaire. For each item, respondents first list the number of individuals available for support in specific circumstances, and then indicate their level of satisfaction with that support using a 6-point Likert-type scale from 1 "dissatisfied" to 6 "very satisfied." The means of the two parts are obtained separately to indicate mean number of social supports and mean satisfaction with social support. The questionnaire will be administered to participants in English by a trained interviewer.
Social support | 6 months
  Participants will complete the 6-item Social Support Questionnaire. For each item, respondents first list the number of individuals available for support in specific circumstances, and then indicate their level of satisfaction with that support using a 6-point Likert-type scale from 1 "dissatisfied" to 6 "very satisfied." The means of the two parts are obtained separately to indicate mean number of social supports and mean satisfaction with social support. The questionnaire will be administered to participants in English by a trained interviewer.
Perceived stress | Baseline
  Participants will complete the Perceived Stress Scale, a 10-item self-report measure that assesses how often a person has experienced thoughts and feelings related to perceived stress over the preceding 1 month. Participants respond on a 5-point Likert scale ranging from 0 "never" to 4 "almost always". Positively worded items are reverse scored, and the responses are summed yielding a score range of 0-40; higher scores indicate more perceived stress. The questionnaire will be administered to participants in English by a trained interviewer.
Perceived stress | 2 months
  Participants will complete the Perceived Stress Scale, a 10-item self-report measure that assesses how often a person has experienced thoughts and feelings related to perceived stress over the preceding 1 month. Participants respond on a 5-point Likert scale ranging from 0 "never" to 4 "almost always". Positively worded items are reverse scored, and the responses are summed yielding a score range of 0-40; higher scores indicate more perceived stress. The questionnaire will be administered to participants in English by a trained interviewer.
Perceived stress | 6 months
  Participants will complete the Perceived Stress Scale, a 10-item self-report measure that assesses how often a person has experienced thoughts and feelings related to perceived stress over the preceding 1 month. Participants respond on a 5-point Likert scale ranging from 0 "never" to 4 "almost always". Positively worded items are reverse scored, and the responses are summed yielding a score range of 0-40; higher scores indicate more perceived stress. The questionnaire will be administered to participants in English by a trained interviewer.
Depressive symptoms | Baseline
  Participants will complete the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short Form, an 8-item self-report measure that assesses depressive symptoms over the preceding 7 days Participants respond on a scale of 1 "never" to 5 "always." Responses are summed to yield a raw score from 8 to 40. Scores may be converted to a T score with score. The questionnaire will be administered to participants in English by a trained interviewer.
Depressive symptoms | 2 months
  Participants will complete the PROMIS Depression Short Form, an 8-item self-report measure that assesses depressive symptoms over the preceding 7 days Participants respond on a scale of 1 "never" to 5 "always." Responses are summed to yield a raw score from 8 to 40. Scores may be converted to a T score with score. The questionnaire will be administered to participants in English by a trained interviewer.
Depressive symptoms | 6 months
  Participants will complete the PROMIS Depression Short Form, an 8-item self-report measure that assesses depressive symptoms over the preceding 7 days Participants respond on a scale of 1 "never" to 5 "always." Responses are summed to yield a raw score from 8 to 40. Scores may be converted to a T score with score. The questionnaire will be administered to participants in English by a trained interviewer.
Anxiety | Baseline
  Participants will complete the PROMIS Anxiety Short Form an 7-item measure about feelings related to anxiety over the preceding 7 days. Participants respond on a 5-point Likert scale from 1 "never" to 5 "always." Responses are summed to yield a raw score from 7 to 35. Scores may be converted to a T score with score. The questionnaire will be administered to participants in English by a trained interviewer.
Anxiety | 2 months
  Participants will complete the PROMIS Anxiety Short Form an 7-item measure about feelings related to anxiety over the preceding 7 days. Participants respond on a 5-point Likert scale from 1 "never" to 5 "always." Responses are summed to yield a raw score from 7 to 35. Scores may be converted to a T score with score. The questionnaire will be administered to participants in English by a trained interviewer.
Anxiety | 6 months
  Participants will complete the PROMIS Anxiety Short Form an 7-item measure about feelings related to anxiety over the preceding 7 days. Participants respond on a 5-point Likert scale from 1 "never" to 5 "always." Responses are summed to yield a raw score from 7 to 35. Scores may be converted to a T score with score. The questionnaire will be administered to participants in English by a trained interviewer.
Type 2 diabetes stigma | Baseline
  Participants will complete the Type 2 Diabetes Stigma Assessment Scale, a 19-item self-report measure assessing domains of being treated differently, blame and judgment, and self-stigma subscales. Participants respond on a 5-point Likert scale from 1 "strongly disagree" to 5 "strongly agree." Item responses are summed to yield subscale and total scores; a higher score indicates presence of more stigma. The questionnaire will be administered to participants in English by a trained interviewer.
Type 2 diabetes stigma | 2 months
  Participants will complete the Type 2 Diabetes Stigma Assessment Scale, a 19-item self-report measure assessing domains of being treated differently, blame and judgment, and self-stigma subscales. Participants respond on a 5-point Likert scale from 1 "strongly disagree" to 5 "strongly agree." Item responses are summed to yield subscale and total scores; a higher score indicates presence of more stigma. The questionnaire will be administered to participants in English by a trained interviewer.
Type 2 diabetes stigma | 6 months
  Participants will complete the Type 2 Diabetes Stigma Assessment Scale, a 19-item self-report measure assessing domains of being treated differently, blame and judgment, and self-stigma subscales. Participants respond on a 5-point Likert scale from 1 "strongly disagree" to 5 "strongly agree." Item responses are summed to yield subscale and total scores; a higher score indicates presence of more stigma. The questionnaire will be administered to participants in English by a trained interviewer.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline A Presley, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Cooper Green Mercy Health Systems, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT05195138/ICF_000.pdf